CLINICAL TRIAL: NCT04549519
Title: Influence of Lumbopelvic Control on Batting Mechanics and Bat-swing Velocity in Baseball Players
Brief Title: Lumbopelvic Control in Baseball Batting
Status: Completed | Type: Observational
Sponsor: National Cheng-Kung University Hospital (Other)
Responsible Party: Principal Investigator, Yi Liang Kuo, Assistant Professor, National Cheng Kung University
Other Study IDs: A-ER-109-197
Record Dates: First submitted 2020-08-23; First posted 2020-09-16 (Actual); Last update posted 2023-11-09 (Actual); Status verified 2023-11

CONDITIONS: Athletes
Keywords: Batting mechanics; Bat-swing velocity; Lumbopelvic control

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Stable group: Participants display knee valgus less or equal to 15° at 45° knee flexion in the descending phase of the squat on both legs
  Interventions: Other: No intervention
- Unstable group: Participants display knee valgus greater than 15° at 45° knee flexion in the descending phase of the squat on one leg or both legs
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention / Compare the difference in batting mechanics and bat-swing velocity in baseball players with good and poor lumbopelvic control

SUMMARY:
Baseball batting is important to winning the games. Baseball batting is achieved by proximal-to-distal sequencing of body movements and controlled by the neuromuscular system. Poor lumbopelvic control could influence production and transfer of energy in the kinetic chain. This study aims to investigate the impact of lumbopelvic control in hitting mechanics and bat swing velocity in high school baseball players.

ELIGIBILITY:
Inclusion Criteria:

* Sport specialization in baseball batting
* Active players on college baseball teams

Exclusion Criteria:

* History of surgery in the lumbar area
* Severe musculoskeletal or neurological symptoms that interfere with participation in competition, training and test

Min Age: 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: College baseball batters in the area of Tainan City
Sampling Method: Non-Probability Sample
Enrollment: 44 (Actual)
Dates: Start 2020-08-17 (Actual); Primary Completion 2022-01-03 (Actual); Study Completion 2022-01-03 (Actual)

PRIMARY OUTCOMES:
Ratio of angular displacement of lumbar spine and hip joint | 1 week after enrolled
  Angular displacement of lumbar spine divided by angular displacement of hip joint
Bat-swing velocity | 1 week after enrolled
  Maximal bat swing velocity during baseball batting
Ratio of angular displacement of thoracic spine and lumbar spine | 1 week after enrolled
  Angular displacement of thoracic spine divided by angular displacement of lumbar spine
Timing of maximal angular velocity of hip joint | 1 week after enrolled
  The time point where the hip joint reaches its maximal angular velocity over the batting phase
Timing of maximal angular velocity of lumbar joint | 1 week after enrolled
  The time point where the lumbar joint reaches its maximal angular velocity over the batting phase
Timing of maximal angular velocity of thoracic joint | 1 week after enrolled
  The time point where the thoracic joint reaches its maximal angular velocity over the batting phase

CONTACTS AND LOCATIONS:
Locations (1):
- National Cheng Kung University, Tainan, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided